CLINICAL TRIAL: NCT05055362
Title: Effect a Honey, Spice-blended Baked Good Has on Salivary Inflammation Markers in Adults: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB202101532
Record Dates: First submitted 2021-09-13; First posted 2021-09-24 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Diseases; Overweight and Obesity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Honey Spice Group (Experimental): The dietary intervention will be a 10-day feasibility trial, using a honey, spice infused baked good. The participants will receive the baked good on day 1 and will be asked to consume a 50-gram baked good daily for 10 days with or without their meals. The honey, spice infused baked good will contain 15g honey and 3g of spice blend (turmeric and cinnamon). A saliva sample will be taken at the start of the intervention (day 1) before consumption of the baked good and after the intervention ends (day 10), 2 hours after consuming the final baked good. Additionally, participants will provide a urine sample to determine microalbuminuria level, complete a spice-consumption survey and a semi-quantitative food frequency questionnaire (day 1). At day 10, participants will indicate if their spice consumption and dietary intake has changed over the past 10 days. Each day, they will tick off the amount of baked good consumed (100%, 75%, 50%, 25%, 0%).
  Interventions: Other: Honey Spice Group

INTERVENTIONS:
Other: Honey Spice Group — Consume baked good daily for 10 days and provide samples of saliva, urine and dietary habits and spice intake.

SUMMARY:
The purpose of this research is to determine the effect a spiced-infused baked good has on inflammatory biomarkers in adults who are overweight and/or who has chronic kidney disease. Participants will be involved for 10 days in this research study.

DETAILED DESCRIPTION:
The dietary intervention will for 10-days, in which participants will eat a baked good each day for a total of 10 days. This baked good contains honey and spices (cinnamon and turmeric). At the first day of the study, participants will provide a urine sample, saliva sample, be weighed, take a pregnancy test, complete a total of 3 surveys - dietary and spice intake and demographics. Each survey will take no more than 10 minutes for a total of 30 minutes. At the end of the 10 days, participants will provide a saliva sample and complete 2 surveys - dietary and spice intake. Each survey will take no more than 10 minutes for a total of 20 minutes. Each day of the baked good intervention, participants will tick off the amount of baked good consumed (100%, 75%, 50%, 25%, 0%).

ELIGIBILITY:
Inclusion Criteria:

* adults who have been diagnosed with CKD and/or have a BMI >24.9
* have no additional chronic diseases or GI disorders or GI disturbances
* age 18 years or older
* no food allergies or dietary restrictions
* all with no contraindications to consuming anything by mouth as per their physician

Exclusion Criteria:

* no diagnosis of CKD or BMI <24.9
* GI disorders, diagnosed with other chronic diseases and conditions, gastrointestinal disturbances
* pregnant and/or lactating
* under 18 years old
* food allergies to wheat, almonds, or aversion to turmeric, cinnamon, and honey. -Dietary restrictions as medically indicated
* trouble chewing/swallowing as confirmed by physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
inflammation markers | 10 days
  Difference in salivary inflammation marker, CRP, concentration pre and post.
inflammation markers | 10 days
  Difference in salivary inflammation marker, IL-6, concentration pre and post.

SECONDARY OUTCOMES:
Dietary and Spice habits | 10 days
  Relationship between dietary and spice habits and inflammation markers

OTHER OUTCOMES:
Albuminuria | 10 days
  Determining relationship between inflammation markers and albuminuria

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Andrade, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Will only be able to provide group information such as demographics